CLINICAL TRIAL: NCT00569751
Title: TAXUS ARRIVE 2: A Multi-Center Safety Surveillance Program
Acronym: ARRIVE 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Kellie Windle, Clinical Project Manager, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2200
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Cardiovascular Disease; de Novo Coronary Lesions
Keywords: de novo; coronary; coronary artery disease; coronary disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: TAXUS™ Express2™ Paclitaxel-Eluting Coronary Stent System — Drug Eluting Stent used to treat de novo coronary artery lesions.

SUMMARY:
The TAXUS ARRIVE 2 study is a multi-center safety and surveillance study designed to to compile safety surveillance and clinical outcomes data for the TAXUS™ Express2™ Paclitaxel-Eluting Coronary Stent System in routine clinical practice and to identify low frequency TAXUS related clinical events.

ELIGIBILITY:
Appropriate Patient Criteria:

* Patient is eligible to receive a Boston Scientific TAXUS Stent

Inappropriate Patient Criteria:

* Known sensitivity to paclitaxel.
* Known allergy to stainless steel.
* Patients in whom antiplatelet and / or anticoagulant therapy is contraindicated.
* Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon or proper placement of the stent or delivery device.
* Patients with unresolved vessel thrombus at the lesion site.
* Patients with coronary artery reference vessel diameters less than 2.5 mm or greater than 3.75 mm.
* Patients with lesions located in the left main coronary artery, ostial lesions, or lesions located at a bifurcation.
* Patients with diffuse disease or poor overflow distal to the identified lesions.
* Patients with tortuous vessels in the region of the obstruction or proximal to the lesion.
* Patients with a recent acute myocardial infarction where there is evidence of thrombus or poor flow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5016 (Actual)
Dates: Start 2004-10; Primary Completion 2006-11 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Rate of TAXUS stent related cardiac events as classified by the Clinical Events Committee (CEC). | 1-year post-implant procedure

SECONDARY OUTCOMES:
Rate of TAXUS stent related cardiac events as classified by the CEC. | within 30 days, 6 months and 2 years
Rate of target vessel related cardiac events as classified by the CEC. | 30 days, at 6 months, at 1 and 2 years post-implant procedure
Rate of other TAXUS related events | 30 days, 6 months, 1 and 2 years post-implant procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Rose, MS, Study Director — Boston Scientific Corporation; John M Lasala, MD, PhD, Principal Investigator — Washington University School of Medicine; David A. Cox, MD, Principal Investigator — Lehigh Valley Physician Group
Locations (53):
- United States (53):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Desert Cardiology Consultants, Rancho Mirage, California
  - Kaiser San Francisco, San Francisco, California
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Health First Clinical Research Institute, Melbourne, Florida
  - Cardiology Consultants, Pensacola, Florida
  - The Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Idaho Cardiology Associates, Boise, Idaho
  - Midwest Heart Foundation, Lombard, Illinois
  - Heart Care Research Foundation, Merrionette Park, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Iowa Heart Center Research, Des Moines, Iowa
  - University of Iowa Hospitals, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - CHRISTUS St. Frances Cabrini Hospital, Alexandria, Louisiana
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Vincent Hospital at Worcester Medical Center, Worcester, Massachusetts
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Great Lakes Heart and Vascular Institute, Saint Joseph, Michigan
  - Minnesota Heart and Vascular Center, Edina, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Barnes / Jewish (Washington University), St Louis, Missouri
  - The Creighton Cardiac Center, Omaha, Nebraska
  - Cardiovascular Associates of Delaware Valley, Haddon Heights, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - Saint Vincent's Catholic Medical Center of New York, New York, New York
  - Mid-Carolina Cardiology Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - HeartCare, Inc, Columbus, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Heart Center of Tulsa, Tulsa, Oklahoma
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Moffitt Heart and Vascular Group, Wormleysburg, Pennsylvania
  - Main Line Health Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Heart Institute, Knoxville, Tennessee
  - St. Thomas Research Institute, Nashville, Tennessee
  - Heart Center of North Texas, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Spectra Clinical Research Management Group, McAllen, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - North Cascade Cardiology, PLLC, Bellingham, Washington
  - Cardiology Associates of Green Bay, Green Bay, Wisconsin
  - South Central Wisconsin Heart, Madison, Wisconsin

REFERENCES:
- [Derived] Brilakis ES, Lasala JM, Cox DA, Berger PB, Bowman TS, Starzyk RM, Dawkins KD. Outcomes after implantation of the TAXUS paclitaxel-eluting stent in saphenous vein graft lesions: results from the ARRIVE (TAXUS Peri-Approval Registry: A Multicenter Safety Surveillance) program. JACC Cardiovasc Interv. 2010 Jul;3(7):742-50. doi: 10.1016/j.jcin.2010.04.012. PMID 20650436
- [Derived] Lasala JM, Cox DA, Dobies D, Baran K, Bachinsky WB, Rogers EW, Breall JA, Lewis DH, Song A, Starzyk RM, Mascioli SR, Dawkins KD, Baim DS; ARRIVE 1 and ARRIVE 2 Participating Physicians. Drug-eluting stent thrombosis in routine clinical practice: two-year outcomes and predictors from the TAXUS ARRIVE registries. Circ Cardiovasc Interv. 2009 Aug;2(4):285-93. doi: 10.1161/CIRCINTERVENTIONS.109.852178.109.852178. Epub 2009 Jul 22. PMID 20031730
- [Derived] Lasala JM, Cox DA, Lewis SJ, Tadros PN, Haas RC, Schweiger MJ, Chhabra A, Untereker WJ, Starzyk RM, Mascioli SR, Dawkins KD, Baim DS. Expanded use of the TAXUS Express Stent: two-year safety insights from the 7,500 patient ARRIVE Registry programme. EuroIntervention. 2009 May;5(1):67-77. doi: 10.4244/eijv5i1a11. PMID 19577985